CLINICAL TRIAL: NCT06527352
Title: Comparison of Risk of Gastroesophageal Reflux During General Anesthesia With Tulip vs GMA(Glottis Mask Airway) Airway
Brief Title: Risk of Gastric Reflux During Tulip vs GMA(Glottis Mask Airway) Airway
Acronym: TUGGER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, Associate professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: XJH-A-20240708
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Anesthesia
Keywords: general anesthesia; glottis mask airway; Tulip shaped tip; gastroesophageal reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- classical shaped mask airway (Other)
  Interventions: Device: glottis mask airway; Other: classical shaped
- tulip shaped mask airway (Other)
  Interventions: Device: glottis mask airway; Other: tulip shaped

INTERVENTIONS:
Device: glottis mask airway — the glottis mask airway is used for maintaining ventilation during general anesthesia
Other: tulip shaped — the tulip shaped mask airway is with a tulip shaped tip
  Arms: tulip shaped mask airway
Other: classical shaped — the classical shaped mask airway is with a water-drop shaped tip
  Arms: classical shaped mask airway

SUMMARY:
Glottis mask airway (GMA) is supraglottic airway device and is frequently used in patients undergoing general anesthesia. However, gastroesophageal reflux remains a risk during ventilation through supraglottic airway devices. The classical shaped GMA and tulip shaped GMA differ in the shape of their tips. And theoretically the tulip shaped tip fits the larynx better. This study aims to compare the incidence of gastroesophageal reflux during ventilation through classical shaped vs tulip shaped glottis mask airway.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years old
* scheduled for surgery under general anesthesia with laryngeal mask airway

Exclusion Criteria:

* American society of anesthesiologists status score higher than 3
* morbid obesity (body mass index higher than 40 kg/m2)
* with high risk of gastroesophageal reflux
* with risk of difficult airway
* with airway disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
pH value of secretion on the tip of glottis mask airway at the end of surgery | at the end of surgery

SECONDARY OUTCOMES:
number of participants with a pH value of secretion on the tip of glottis mask airway less than 4.1 | at the end of surgery
Oropharyngeal leak pressure | from insertion of glottis mask airway to start of surgery, at an average of 10 minutes
  Oropharyngeal leak pressure (OLP) was measured by setting the adjustable pressure limiting valve to 40 cmH2O at a fixed gas flow of 3 L/min and noting the steady-state airway pressure on the monitor
duration of inserting glottis mask airway | from taking of glottis mask airway to inserting it to appropriate position, at an average of 1 minute
number of insertion to achieve successful positioning of glottis mask airway | from taking of glottis mask airway to inserting it to appropriate position, at an average of 1 minute
duration of establishing appropriate ventilation | from taking of glottis mask airway to inserting it to appropriate position, at an average of 1 minute
incidence of epiglottis suppression | from insertion of glottis mask airway to start of surgery, at an average of 10 minutes
number of needs for modulating the position of glottis airway mask during surgery | from insertion of glottis mask airway to end of surgery, at an average of 2 hours
scale of difficulty of inserting gastric tube | from insertion of glottis mask airway to start of surgery, at an average of 10 minutes
  0 is for easy to insert; 1 is for a little difficult to insert; 2 is for fail to insert
incidence of blood on the tip of glottis airway mask | from end of surgery to withdrawal of glottis airway mask, at an average of 5 minutes
score of satisfaction of anesthesiologist to glottis airway mask | from insertion of glottis mask airway to withdrawal of glottis airway mask, at an average of 2 hours
  the score is from 0 to 10, a higher score means higher satisfaction
incidence of glottis airway mask related adverse events by 24 hours after surgery | 24 hours after surgery
  the glottis airway mask related adverse events include laryngeal pain, horse and dysphonia

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Air Force Medical University, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Lemos J, De Oliveira GS Jr, de Pereira Cardoso HE, Lemos LD, de Carvalho LR, Modolo NS. Gastric regurgitation in patients undergoing gynecological laparoscopy with a laryngeal mask airway: a prospective observational study. J Clin Anesth. 2017 Feb;36:32-35. doi: 10.1016/j.jclinane.2016.07.038. Epub 2016 Nov 11. PMID 28183569
- [Background] Nakanishi T, Sakamoto S, Yoshimura M, Toriumi T. AutoFlow(R) versus volume-controlled ventilation for laparoscopic gynecological surgery using LMA(R) ProSeal: a randomized controlled trial. BMC Anesthesiol. 2021 Jun 28;21(1):181. doi: 10.1186/s12871-021-01406-6. PMID 34182933
- [Result] Liu Y, Song Y, Wang M, Yang M, Shen H, Wang Z, Chen L, Yang J, Gong S, Yu Y, Shi Z, Zhang W, Zou X, Sun X, Wang Y, Fu Q, Cao J, Mi W. LMA(R) protector in patients undergoing laparoscopic surgeries: a multicenter prospective observational study. BMC Anesthesiol. 2021 Dec 20;21(1):318. doi: 10.1186/s12871-021-01535-y. PMID 34930137
- [Result] Bhardwaj M, Dhania S, Kaur K, Lal J, Priya, Singhal SK. Comparison of oropharyngeal leak pressure of LMA Protector and LMA ProSeal in anaesthetised paralysed patients - A randomised controlled trial. Indian J Anaesth. 2023 Nov;67(Suppl 4):S245-S250. doi: 10.4103/ija.ija_403_23. Epub 2023 Nov 21. PMID 38187973